CLINICAL TRIAL: NCT05468073
Title: Therapeutic Evaluation of Low-dose IL-2-based Immunomodulatory Approach in Patients With Early AD
Acronym: IL-2-AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: For Drug Consulting (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D20-P012
Record Dates: First submitted 2020-12-21; First posted 2022-07-21 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: Interleukin; Neuroinflammation; Regulatory T cells; Microglia; Synaptic density
MeSH Terms: conditions — Alzheimer Disease; Neuroinflammatory Diseases | interventions — aldesleukin; Interleukin-2; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patient will be treated with low dose of Interleukin 2 (PROLEUKIN ®)
  Interventions: Drug: Proleukin
- Placebo (Placebo Comparator): Patient will receive sodium chloride solution (NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proleukin — Sub-cutaneous injections of Interleukin-2 (PROLEUKIN ®) Induction phase: 5 consecutive days. A week break. Maintenance phase: once a week during 16 weeks
  Other Names: Interleukin 2
  Arms: Treatment
Drug: Placebo — Sub-cutaneous injections of placebo (NaCl) Induction phase: 5 consecutive days. A week break. Maintenance phase: once a week during 16 weeks.
  Other Names: Sodium chloride solution
  Arms: Placebo

SUMMARY:
Study aims at evaluating the therapeutic efficacy and safety of low-dose IL-2 immunomodulatory treatment in patients with early AD, in a phase II, randomized, double blind, placebo-controlled phase II clinical trial. Patients with AD at early stage will be recruited and randomized (2:1) in each treatment group.

The primary endpoint is the rate of decline assessed through CDR change at 18 months between the placebo group and the treated patients.

DETAILED DESCRIPTION:
This study aims to investigate the immunomodulatory therapeutic potential and safety of low-dose (ld) IL-2 in a randomized, double blind, and placebo-controlled phase II clinical trial.

Conservative diagnosis criteria based on clinical and CSF biomarkers have been established to avoid risks of misdiagnosis.

The treatment consist of 21 cures of subcutaneous injections of either placebo or low-dose (1MIU/day) IL-2 (PROLEUKIN ®). Patients will receive 5 consecutive injections during the induction phase which will be followed by a week break. During the maintenance phase a total of 16 injections will be administered weekly. Total duration of treatment for each patient is anticipated to be 18 weeks. Patients will be followed-up for 18 months after the first injection.

At inclusion, in addition to the clinical evaluation, a hybrid PET/MRI (using [18F]-DPA-714) scan will be performed. After randomized patients successfully complete the treatment phases, they will be followed-up through 3 clinical and 1 neuroimaging visits to assess cogitive and functional decline. Clinical visits are scheduled at 6, 12, and 18 months after treatment induction. Another hybrid PET/MRI (using [18F]-DPA-714) scan will be performed at 19 months following induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18
* Age of disease onset < 70 years
* Clinical and biological diagnosis of AD based on

  * Progressive amnestic syndrome associated or not with other cognitive impairments
  * Biological criteria: CSF biomarkers suggestive of AD.
* Brain MRI congruent with the diagnosis, left to the appreciation of the investigator
* CDR (Clinical Dementia Rating Scale) = 0.5 or 1
* If patients have an antidepressant or acetylcholinesterase inhibitors treatment, patients must be treated with stable doses of treatment for at least 1 month before inclusion.
* Have a caregiver who provides a separate written informed consent to participate. If a caregiver/study informant cannot continue, one replacement is allowed.
* Have adequate vision and hearing for neuropsychological testing in the opinion of the investigator.
* Have given written informed consent approved by the ethical review board (ERB) governing the site.
* The patient has to have a French social security number and be fluent and literate in French.

Exclusion Criteria:

* Subject with a psychiatric evolutionary and/or badly checked.
* Subject with a grave, severe or unstable pathology (left to the judgement of the investigator) the nature of which can interfere with the variables of evaluation.
* Epileptic subjects
* Subject under guardianship or curatorship
* Subject presenting contraindications to the MRI
* Known or supposed history (< or = 5 years) of severe alcoholism or misuse of drugs
* Vascular, inflammatory or expansive, visible lesion in the MRI, which can interfere on the criteria of diagnosis.
* No health insurance
* Women of childbearing potential: a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* History of auto-immune disease
* History within the past 10 years of a primary or recurrent malignant disease
* Diagnosis or history of other possible etiology of dementia, including but not limited to other neurodegenerative disorders (FTD, LBD, VaD, HD, PD, PSP-CBD).
* Renal dysfunction at inclusion, clearance <30 mL/min
* Chronic hepatic diseases as indicated by liver function tests abnormalities
* Abnormal thyroid function
* Therapeutic trial within 1 year preceding the first study period, or participation in a trial with active or passive immunization against amyloid if patient was assigned to the active treatment arm.
* Clinically significant evidence of Active viral infection (CMV, EBV, HCV, HBV, TPHA-VDRL, HIV)
* Current or medical history of severe cardiopathy,
* - Severe dysfunction in a vital organ
* Patients with White Blood Count (WBC) < 4.000/mm3; platelets < 100.000/mm3; hematocrit (HCT) < 30%.
* Patients with serum bilirubin and creatinine outside normal range.
* Patients with organ allografts.
* Patients who are likely to require corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline CDR score at 18 months | 18 months
  The primary endpoint will be evaluated in all patients evaluable for efficacy, i.e. patients who received at least one cure of IL-2 and were evaluated for cognitive and functional status at baseline and 18 months.
  The response variable will be dichotomized as follows:
  Responder patient = 1 (end of study CDR score <= baseline CDR score)
  Non-responder patient = 0 (end of study CDR score > baseline CDR score)

SECONDARY OUTCOMES:
Rate of cognitive decline between placebo and treatment groups as assessed by changes in MMSE scores at baseline, 6, 12, and 18 months | 6, 12 and 18 months
  MMSE total score out of 30
Rate of cognitive decline between placebo and treatment groups as assessed by changes in ADAS-Cog 13 items scores at baseline, 6, 12, and 18 months | 6, 12 and 18 months
  ADAS-Cog total score out of 85
Rate of functional decline between placebo and treatment groups as assessed by changes in ADCS-ADL MCI scores at baseline, 6, 12, and 18 months | 6, 12 and 18 months
  ADSC-ADL MCI total score out of 53
Rate of functional decline between placebo and treatment groups as assessed by changes in CDR (sum of boxes) scores at baseline, 6, 12, and 18 months | 6, 12 and 18 months
  CDR sum of the boxes (CDR-SOB) total score out of 18
Change in neuroimmune reaction as assessed by [18F]-DPA-714 PET global cortical index and regional cortical binding at baseline and 18 months between placebo and treated groups | 18 months
  Global and regional cortical [18F]-DPA-714 PET uptake ratio
Change in peripheral frequency of Treg and other immune effectors at 18 months compared to baseline between placebo and treated groups | 6, 12 and 18 month
  Tregs frequency, total lymphocytes as a biomarker of target engagement
Change in hippocampal atrophy at 18 month compared to baseline between placebo and treated groups | 18 months
  Volume of hippocampus measured in T1 MRI
Number of patients with treatment related adverse events as assessed by clinical safety panel | 18 months
  Clinical safety will be assessed via the following assessments:
  Vital signs (including blood pressure, weight, BPM, temperature) - each visit
  ECG - at inclusion and at V22 (M18)
  Check-list questionnaire to assess clinical adverse events - each visit
Number of patients with treatment related adverse events as assessed by blood laboratory safety panel | 18 months
  Biological safety will be evaluated and controlled through blood laboratory safety tests which include the following:
  Thyroid function: T4 and TSH - at inclusion, at V21
  Haematology (RBC, WBC, leukocyte formula, platelets) and C reactive protein (CRP) - at inclusion, 8 days before the randomization, each day of the induction phase (day 1 to day 5), before each injection of the maintenance phase until V7, then every fortnight until the last injection of the maintenance phase, and then at M6, M12 and M18.
  Biochemistry (electrolytes, proteins, albumin, urea, creatinine, glucose, AST, ALT, GGT, bilirubin) and Coagulation tests - at inclusion, 8 days before the randomization, every 2 months for 6 months (V9 and V17), and at M6, M12 and M18

CONTACTS AND LOCATIONS:
Overall Officials: Marie SARAZIN, Prof, Principal Investigator — GHU Saint Anne; Guillaume DOROTHEE, PhD, Study Chair — INSERM UMRS 938; Michel BOTTLAENDER, Dr, Study Chair — Service Hospitalier Frédéric Joliot / CEA
Locations (1):
- GHU Saint Anne, Paris, France

IPD SHARING:
Plan to Share IPD: No